CLINICAL TRIAL: NCT00002256
Title: Dideoxycytidine ( Ro 24-2027 ). A Treatment Protocol for the Use of Dideoxycytidine ( ddC ) in Patients With AIDS or Advanced ARC Who Cannot Be Maintained on Zidovudine ( AZT ) Therapy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 031D; N3663
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-08

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zalcitabine

INTERVENTIONS:
Drug: Zalcitabine

SUMMARY:
To provide zalcitabine ( ddC ) for patients with AIDS or Advanced ARC in whom zidovudine ( AZT ) is contraindicated, or who have failed treatment with or are intolerant to AZT and to demonstrate that ddC monotherapy is safe, and tolerable in this patient population.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized Pentamidine or Trimethoprim/sulfamethoxazole prophylaxis against Pneumocystis carinii pneumonia is recommended.
* Dapsone is permitted but discouraged.
* Drugs that could cause other serious toxicity when coadministered with study medication is allowed for treatment of an acute intercurrent illness or opportunistic infection at the investigator's discretion.
* Any medication that has the potential to cause peripheral neuropathy should be avoided; patients should consult their physicians for specific drugs.
* Isoniazid is permitted if there is no evidence of peripheral neuropathy at entry and the patient is taking pyridoxine = or > 50 mg/day.
* Metronidazole is permitted only with a study drug interruption.
* Patients on amphotericin, pyrimethamine, sulfadiazine, trimethoprim/sulfamethoxazole, ganciclovir, intravenous pentamidine, intravenous acyclovir = or > 1000 mg/day orally or other bone marrow or renal toxic drugs may not tolerate concomitant ddC. If these drugs are given concomitantly with ddC, patients should have frequent (weekly) laboratory assessments, as appropriate.
* Drugs that are nephrotoxic or have the potential to cause peripheral neuropathy might be expected to cause increased toxicity when co-administered with ddC.
* The following experimental medications are allowed if, in the judgement of the investigator, no serious additive toxicities are anticipated and the experimental drug is necessary for optimal patient management:
* Ampligen, azithromycin, BW 566C80, bovine colostrum, clarithromycin, diclazuril, foscarnet, oral ganciclovir, GM-CSF, G-CSF, hypericin, IL-2, interferon-beta, interferon-gamma, itraconazole, liposomal amphotericin, liposomal gentamicin, nimodipine, PEG-IL2 (polyethylene glycosylated IL-2), roxithromycin, spiramycin, trimetrexate.

Patients must have the following:

* AIDS or Advanced ARC.
* Patients eligible to enter this protocol must fall into one of the following three categories:
* AZT treatment failure or AZT intolerance or AZT ineligibility or Rollover Patients Under 18 years of age must have the consent of a parent or guardian.

Exclusion Criteria

Patients with the following are excluded:

* Any history of peripheral neuropathy due to any cause, even if peripheral neuropathy was not the reason for discontinuation of other anti-HIV therapy.
* Any finding suggestive of peripheral neuropathy found at baseline neurological exam. If a patient has an isolated finding of an absent achilles reflex he may be entered if no signs or symptoms and no other findings are suggestive of peripheral neuropathy.
* Concomitant treatment with excluded medications. Excluded medications include any other experimental drugs (including ddI), drugs with known nephrotoxic or hepatotoxic potential, and drugs likely to cause peripheral neuropathy. Any = or > Grade 3 laboratory or clinical abnormality or any severe abnormality not listed requires permission from the medical monitor to be entered into this study..
* Unwillingness or deemed unable to sign informed consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Hoffmann - La Roche Inc, Nutley, New Jersey, United States